CLINICAL TRIAL: NCT05992363
Title: Tandem Polyurethane Stents Compared to Single Silicone Stent for Malignant Ureteral Obstruction
Acronym: TSTENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Michael Frumer, Urologist, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0100-23-RMC
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Hydronephrosis; Obstruction, Ureter; Renal Failure; Malignancy; Ureter Obstruction; Ureter Stricture
MeSH Terms: conditions — Hydronephrosis; Bites and Stings; Renal Insufficiency; Neoplasms; Ureteral Obstruction

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- single silicone stent (Active Comparator): patients with malignant ureteral obstruction that was treated by single large-caliber 8-12Fr silicone stent
  Interventions: Device: ureteral stent\s insertion
- Tandem polyurethane stents (Active Comparator): patients with malignant ureteral obstruction that was treated by tandem 6 Fr Percuflex™ stents
  Interventions: Device: ureteral stent\s insertion

INTERVENTIONS:
Device: ureteral stent\s insertion — ureteral stent\s insertion in the operating room

SUMMARY:
Malignant ureteral obstruction (MUO) is an extrinsic ureteral obstruction caused by malignant diseases. This study aim to compare tandem 6 Fr Percuflex™ stents and single large-caliber 8Fr silicone stent in patients with MUO. The primary endpoint is stent failure rate. The secondary endpoints are patient comfort, quality of life and overall survival.

DETAILED DESCRIPTION:
Malignant ureteral obstruction (MUO) is an extrinsic ureteral obstruction caused by malignant diseases. MUO may induce renal failure, which would be a barrier to several therapies including chemotherapy. Indwelling double-pigtail polymeric ureteral stent is a common method to release renal obstruction, but does not necessarily guarantee renal decompression as most studies reported stent failure with a mean of 30% at a mean time of three months [1-3]. Various endoscopic strategies have been proposed to increase time to failure, including tandem polymeric stents, metallic spiral coil stent, self-expanding Nitinol stent and polymeric stents with different lumen diameter and stiffness [4-7]. However, heterogeneity of MUO, low number of patients, unspecified polymer type, retrospective studies and the lack of a standard method to assess stent failure limit robust comparative analysis.

Tandem ureteral stents (TUS) technique uses two polymeric ureteral stents passed simultaneously to better withstand the presumed compressive forces that overcome conventional single stent. This method offers an additional parallel lumen and allows more extraluminal flow between the two stents [6].

In a study on TUS in 39 renal units with MUO, two 6 Fr stents were inserted. Stent failure, defined by flank pain with increasing creatinine level or worsening hydronephrosis during 3 months after stents insertion, was occurred in 4% of cases [7]. This low failure rate compares favorably with the reported rates with single 6Fr polymeric stent or metallic stent. However, stents irritation, defined by profound lower urinary tract symptoms or renal colic in the absence of worsening hydronephrosis or infection, was reported in 29-85% of patients [7,8].

Silicon stent, which is considered biocompatible and soft, has the potential to be less irritative. In a recent systematic review, silicone stents has less stent-related symptoms in comparison to non-silicone polymers and ''hard'' stents. [9]. However, silicone has high susceptibility to compression, which in case of MUO may results in lower drainage efficacy.

This study aim to compare tandem 6 Fr Percuflex™ stents and single large-caliber 8Fr silicone stent in patients with MUO. The primary endpoint is stent failure rate. The secondary endpoints are patient comfort, quality of life and overall survival.

References:

1. Docimo SG, Dewolf WC. High failure rate of indwelling ureteral stents in patients with extrinsic obstruction: experience at 2 institutions. J Urol. 1989;142(2 Pt 1):277-279. doi:10.1016/s0022-5347(17)38729-3
2. Vogt B, Blanchet LH. Analysis of Ureteral Tumour Stents for Malignant Ureteral Obstruction: Towards Reshaping an Optimal Stent. Res Rep Urol. 2021;13:773-782. Published 2021 Oct 27. doi:10.2147/RRU.S334277
3. Chung SY, Stein RJ, Landsittel D, et al. 15-year experience with the management of extrinsic ureteral obstruction with indwelling ureteral stents. J Urol. 2004;172(2):592-595. doi:10.1097/01.ju.0000130510.28768.f5
4. Patel C, Loughran D, Jones R, Abdulmajed M, Shergill I. The resonance® metallic ureteric stent in the treatment of chronic ureteric obstruction: a safety and efficacy analysis from a contemporary clinical series. BMC Urol. 2017;17(1):16. Published 2017 Mar 10. doi:10.1186/s12894-017-0204-8
5. Khoo CC, Ho C, Palaniappan V, et al. Single-Center Experience with Three Metallic Ureteral Stents (Allium® URS, Memokath™-051, and Resonance®) for Chronic Ureteral Obstruction. J Endourol. 2021;35(12):1829-1837. doi:10.1089/end.2021.0208
6. Fromer DL, Shabsigh A, Benson MC, Gupta M. Simultaneous multiple double pigtail stents for malignant ureteral obstruction. Urology. 2002;59(4):594-596. doi:10.1016/s0090-4295(01)01646-7
7. Elsamra SE, Motato H, Moreira DM, et al. Tandem ureteral stents for the decompression of malignant and benign obstructive uropathy. J Endourol. 2013;27(10):1297-1302. doi:10.1089/end.2013.0281
8. Shvero A, Haifler M, Mahmud H, Dotan Z, Winkler H, Kleinmann N. Quality of life with tandem ureteral stents compared to percutaneous nephrostomy for malignant ureteral obstruction. Support Care Cancer. 2022;30(11):9541-9548. doi:10.1007/s00520-022-07354-2
9. Boeykens M, Keller EX, Bosio A, et al. Impact of Ureteral Stent Material on Stent-related Symptoms: A Systematic Review of the Literature. Eur Urol Open Sci. 2022;45:108-117. Published 2022 Oct 19. doi:10.1016/j.euros.2022.09.005

ELIGIBILITY:
Inclusion Criteria:

* patient with malignant ureteral obstruction

Exclusion Criteria:

* ureteral obstruction of other causes
* Language comprehension or other limitation in giving informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
stent failure rate | 1 year
  Failure will be defined when two of the following three appear: renal colic, rise in serum creatinine, hydronephrosis

SECONDARY OUTCOMES:
quality of life score | 1 year
  using the Ureteral stent symptom questionnaire (USSQ) score
overall survival | 1 year
  overall survival

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Rabin Medical Center, Petah Tikva
  - Sheba medical center, Ramat Gan

IPD SHARING:
Plan to Share IPD: No